CLINICAL TRIAL: NCT01479114
Title: In Vivo Effect of Recombinant Human Granulocyte Colony- Stimulating Factor on Neutrophilic Expression of CD11b in Septic Neonates
Brief Title: Effect of Recombinant Human Granulocyte Colony- Stimulating Factor on CD11b in Septic Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC 09030
Record Dates: First submitted 2011-11-21; First posted 2011-11-24 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (No Intervention)
- G-CSF group (Experimental)
  Interventions: Drug: rh-GCSF
- Non-GCSF group (No Intervention)

INTERVENTIONS:
Drug: rh-GCSF — 10 ug/kg/day intravenously for 3 days
  Other Names: Granulocyte colony stimulating factor,neubogen,filgstrim
  Arms: G-CSF group

SUMMARY:
The investigators aimed to evaluate the effect of G-CSF administration in septic neonates on neutrophil production and CD11b expression.

DETAILED DESCRIPTION:
Neonates are susceptible to septicemia secondary to quantitative and qualitative neutrophilic defects. Granulocyte-colony stimulating factor (G-CSF) stimulates myeloid progenitor cell proliferation and induces selective neutrophil functions.

ELIGIBILITY:
Inclusion Criteria:

* newborn infants with postnatal age < 28 day,
* minimum gestational age of 28 weeks and requiring intensive care with clinical signs consistent with the diagnosis of neonatal sepsis,
* with or without neutropenia

Exclusion Criteria:

* neonates with congenital malformation,
* major chromosomal abnormalities,
* prior use of cytokines or intravenous immunoglobulin, or decreased hemoglobin and/or hematocrit at or below the levels necessitate transfusion

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one month